CLINICAL TRIAL: NCT04893915
Title: A Phase 2 Study of Cytokine-induced Memory-like NK Cells in Relapsed/Refractory AML and MDS
Brief Title: Cytokine-induced Memory-like NK Cells in Relapsed/Refractory AML and MDS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding support
Sponsor: Washington University School of Medicine (Other)
Collaborators: Wugen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202106075
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — fludarabine; Cyclophosphamide; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lead In Cohort Recipient: Cytokine-induced memory-like NK cells (Experimental): * Fludarabine and cyclophosphamide beginning on Day -6.
  * NK cell product will be infused on Day 0.
  * IL-2 will begin 2-4 hours after infusion and will continue every other day through Day 12 for a total of 7 doses.
  * NK cell product will be infused into the recipient on Day +14.
  * IL-2 will begin 2-4 hours after infusion and will continue every other day through Day 26 for an additional 7 doses, and a total of 14 doses, to a maximum of two vials of rhIL-2 per IL-2 course.
  * In the Lead-in Cohort, three patients will receive NK cell product on Day 0 and Day +14, receiving the maximum NK cells generated, capped at 20x10^6/kg.
  * Patients that have an initial response but then subsequently relapse or progress will be able to receive a third dose of NK cell product with or without lymphodepleting chemotherapy depending on the interval duration between the second dose and relapse, after approval by the study PI. The third dose should be administered not less than 45 days from Day 0.
  Interventions: Biological: Cytokine-induced memory-like NK cells; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Interleukin-2
- Phase II Recipient: Cytokine-induced memory-like NK cells (Experimental): * Fludarabine and cyclophosphamide beginning on Day -6.
  * NK cell product will be infused on Day 0.
  * IL-2 will begin 2-4 hours after infusion and will continue every other day through Day 12 for a total of 7 doses.
  * NK cell product will be infused into the recipient on Day +14.
  * IL-2 will begin 2-4 hours after infusion and will continue every other day through Day 26 for an additional 7 doses, and a total of 14 doses, to a maximum of two vials of rhIL-2 per IL-2 course.
  * Will receive the NK cell product on Day 0 and Day +14, receiving the maximum NK cells generated, capped at 20x10^6/kg.
  * Patients that have an initial response but then subsequently relapse or progress will be able to receive a third dose of NK cell product with or without lymphodepleting chemotherapy depending on the interval duration between the second dose and relapse, after approval by the study PI. The third dose should be administered not less than 45 days from Day 0.
  Interventions: Biological: Cytokine-induced memory-like NK cells; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Interleukin-2
- Donor (Experimental): * The allogeneic donor will undergo non-mobilized large volume (20-L) leukapheresis on Day -1.
  * On Day +13 the allogeneic donor will again undergo non-mobilized large volume (20-L) leukapheresis
  Interventions: Procedure: Donor Leukapheresis

INTERVENTIONS:
Biological: Cytokine-induced memory-like NK cells — Cell product processing is performed at the Siteman Cancer Center Biological Therapy Core or another FACT-accredited cellular therapy production facility that can manufacture the product per the IND CMC.
  Arms: Lead In Cohort Recipient: Cytokine-induced memory-like NK cells; Phase II Recipient: Cytokine-induced memory-like NK cells
Drug: Fludarabine — -Lymphodepleting regimen
  Arms: Lead In Cohort Recipient: Cytokine-induced memory-like NK cells; Phase II Recipient: Cytokine-induced memory-like NK cells
Drug: Cyclophosphamide — -Lymphodepleting regimen
  Arms: Lead In Cohort Recipient: Cytokine-induced memory-like NK cells; Phase II Recipient: Cytokine-induced memory-like NK cells
Procedure: Donor Leukapheresis — -Apheresis will be performed via peripheral IVs or central line, as determined by the apheresis team.
  Arms: Donor
Drug: Interleukin-2 — -IL-2 will start approximately 2-4 hours after the NK cell infusions.
  Other Names: IL-2
  Arms: Lead In Cohort Recipient: Cytokine-induced memory-like NK cells; Phase II Recipient: Cytokine-induced memory-like NK cells

SUMMARY:
Patients with relapsed/refractory acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) will receive lymphodepleting chemotherapy (Flu/Cy) and two infusions of cytokine-induced memory-like NK cells at the previously defined maximum tolerated dose (MTD), fourteen days apart. Low dose rhIL-2 will be administered to patients for in vivo expansion following cell infusion. Patients will be assessed for anti-leukemic efficacy and safety. Re-infusion of patients who relapsed after clinical response will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Refractory AML without CR after induction therapy (primary induction failure); relapsed AML after obtaining a CR; progressive AML after non-intensive therapy (e.g., HMA + venetoclax or targeted therapy); Intermediate risk to very-high-risk MDS by IPSS-R that is relapsed or refractory after prior therapy with an HMA-containing regimen
* At least 18 years of age.
* Available allogeneic donor that meets the following criteria:

  * Able and willing to undergo multiple rounds of leukapheresis
  * At least 18 years of age
  * In general good health, and medically able to tolerate leukapheresis required for harvesting the NK cells for this study.
  * Negative for hepatitis, HTLV, and HIV on donor viral screen
  * Not pregnant
  * Voluntary written consent to participate in this study
  * All HLA-match/mismatch statuses will be included, with preference for unmatched donors all else being equal
* Patients with known CNS involvement with AML are eligible provided that they have been treated and CSF is clear for at least 2 weeks prior to enrollment into the study. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the study treatment.
* Karnofsky/Lansky performance status > 50 %
* Adequate organ function as defined below:

  * Total bilirubin < 2 mg/dL
  * AST(SGOT)/ALT(SGPT) < 3.0 x ULN
  * Creatinine within normal institutional limits OR creatinine clearance ≥ 40 mL/min by Cockcroft-Gault Formula
  * Oxygen saturation ≥90% on room air
  * Ejection fraction ≥35%
* Able to be off corticosteroids and any other immune suppressive medications beginning on Day -3 and continuing until 30 days after the last infusion of the NK cell product. However, use of low-level corticosteroids is permitted if deemed medically necessary. Low-level corticosteroid use is defined as 10mg or less of prednisone (or equivalent for other steroids) per day.
* Women of childbearing potential must have a negative pregnancy test within 28 days prior to study registration. Female and male patients (along with their female partners) must agree to use two forms of acceptable contraception, including one barrier method, during participation in the study and until 30 days after the last NK cell product infusion.
* Ability to understand and willingness to sign an IRB approved written informed consent document

Exclusion Criteria:

* Relapsed after allogeneic transplantation.
* Circulating blast count >30,000/µL by morphology or flow cytometry (cytoreductive therapies including leukapheresis or hydroxyurea are allowed).
* Uncontrolled bacterial or viral infections, or known HIV, Hepatitis B or C infection.
* Uncontrolled angina, severe uncontrolled ventricular arrhythmias, or EKG suggestive of acute ischemia or active conduction system abnormalities.
* New progressive pulmonary infiltrates on screening chest x-ray or chest CT scan that have not been evaluated with bronchoscopy. Infiltrates attributed to infection must be stable/ improving after 1 week of appropriate therapy (4 weeks for presumed or proven fungal infections).
* Known hypersensitivity to one or more of the study agents.
* Received any investigational drugs within the 14 days prior to the first dose of fludarabine.
* Pregnant and/or breastfeeding.
* Any condition that, in the opinion of the investigator, would prevent the participant from consenting to or participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) of recipients | Through 12 month follow-up
  * Defined as the proportion of patients achieving complete remission (CR), complete remission with partial hematologic recovery (CRh), and complete remission with incomplete blood count recovery (CRi).
  * Response will be assessed according to the criteria from the International Working Group Response Criteria

SECONDARY OUTCOMES:
Overall survival (OS) of recipients | Through completion of follow-up (estimated to be 12 months)
  -Defined as time from first dose of lymphodepleting chemotherapy (LDC) until death from any cause
Event free survival (EFS) of recipients | Through completion of follow-up (estimated to be 12 months)
  -Defined as time from first dose of lymphodepleting chemotherapy (LDC) until treatment failure, relapse from complete response, or death
Duration of overall response (DOR) of recipients | Through 12 month follow-up
  -Defined as duration for first occurrence of documented ORR until disease progression or death
Duration of complete response (DoCR) of recipients | Through 12 month follow-up
  -Defined as duration from documented complete remission until disease progression or death
Proportion of recipients that receive multiple doses of NK cell product | Through Day +14 of all recipients enrolled (estimated to be 19 months)
Number of dose-limiting toxicities (DLTs) that recipients experience in the safety lead-in cohort | Through Day 28
Mortality rate of recipients | Day +30
Mortality rate of recipients | Day +100
Number of adverse events experienced by recipients | Through Day +100
  * Incidence, nature, and severity of adverse events
  * Adverse events will be collected from Day 0 to Day +35; however, bone marrow suppression (ANC < 500/µL) and adverse events of graft-versus-host disease (GVHD) involving the liver, skin, or gastrointestinal tract will be recorded until Day +100.
Proportion of recipients with prolonged cytopenia | At 8 weeks
Change in quality of life experienced by recipients as measured by the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire (EORTC QLQ-C30) | Day 0, Day +28, Day +100, 6 months, 9 months, and 12 months
Overall response rate (ORR) of recipients compared across subgroups | Through 12 month follow-up
  * Subgroups will be defined by degree of HLA-match from allogeneic donor
  * Defined as the proportion of patients achieving complete remission (CR), complete remission with partial hematologic recovery (CRh), and complete remission with incomplete blood count recovery (CRi).
  * Response will be assessed according to the criteria from the International Working Group Response Criteria
Number of adverse events experienced by recipients compared across subgroups | Through Day +100
  * Subgroups will be defined by degree of HLA-match from allogeneic donor
  * Incidence, nature, and severity of adverse events
  * Adverse events will be collected from Day 0 to Day +35; however, bone marrow suppression (ANC < 500/µL) and adverse events of graft-versus-host disease (GVHD) involving the liver, skin, or gastrointestinal tract will be recorded until Day +100.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cashen, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu